CLINICAL TRIAL: NCT04965441
Title: Computer-assisted Versus Traditional Freehand Technique for Mandibular Reconstruction With Free Vascularized Fibular Flap: A Matched-pair Study
Brief Title: CAS Versus Traditional Freehand Technique for Mandibular Reconstruction With Free Vascularized Fibular Flap
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Hongyang Ma, Principal Investigator, KU Leuven
Other Study IDs: S63615-2
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Operation Time; Complication of Surgical Procedure
Keywords: Computer-Assisted Surgeries; Mandibular Reconstruction; Matched-Pair Analysis
MeSH Terms: interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Computer-assisted surgery (CAS) group
  Interventions: Procedure: Computer-assisted surgery
- Non-CAS group

INTERVENTIONS:
Procedure: Computer-assisted surgery — Preoperative head and neck computed tomography (CT) and lower extremity CT angiography were acquired for all patients. In the CAS group, CT images (slice thickness<1 mm) were imported into a 3D surgical planning software (Proplan, Version 2.0/3.0 Materialise, Leuven, Belgium). Virtual surgical planning was performed to determine the mandibular and fibular resection and cut margins with localization of the optimal angles for performing osteotomies. After that, surgical guides were designed utilizing a 3D designing software (3-Matic, Version 9.0-13.0, Materialise, Leuven, Belgium). The generated virtual templates were exported in Standard Tessellation Language (STL) format and printed with a professional 3D printer (Connex 350, Stratasys, Eden Prairie, MN, USA). The reconstructive plates were pre-bent on a 3D printed planned mandibular model.
  Groups: Computer-assisted surgery (CAS) group

SUMMARY:
A total of 153 patients who underwent mandibular reconstruction by VFF were included from Jan 1999 to Dec 2019. The mandibular resection and reconstruction were performed by four experienced oral and maxillofacial surgeons. Reasons for reconstruction were oncologic, osteoradionecrosis, trauma, and osteoporosis. All the patients were followed up postoperatively for at least one year. Eighteen pairs were formed with the matched cohort consisting of a total of 36 patients who underwent primary mandibular reconstruction without additional combined flaps. The surgery-related and patient-related continuous and categorical parameters were assessed in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of head and neck cancer
* Received mandibular reconstruction
* All patients were followed up postoperatively for at least one year

Exclusion Criteria:

* Patients received bone graft for jaw reconstruction before mandibular reconstruction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 153 patients who underwent mandibular reconstruction by VFF were included from Jan 1999 to Dec 2019.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
operation time | within the surgery
  operation time

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No